CLINICAL TRIAL: NCT06285968
Title: Addressing Sleep Duration, Regularity, and Efficiency: A Multidimensional Sleep Health Intervention for Improving Cardiometabolic Health (The DREAM Study)
Brief Title: The DREAM Study: A Multidimensional Sleep Health Intervention for Improving Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Nour Makarem, PhD, Assistant Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAU8937; P50MD017341 (NIH)
Record Dates: First submitted 2024-02-13; First posted 2024-02-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidimensional Sleep Health Promotion Intervention (Experimental): Participants randomized to the intervention arm will receive:
  1. A multi-component multidimensional sleep health promotion intervention that includes report back of sleep health profiles, S.M.A.R.T. goal setting, sleep health coaching, establishment of fixed sleep schedule, virtual sleep hygiene education, self-monitoring, personalized feedback and supportive accountability, and addressing light and noise in the sleep environment.
  2. Cardiovascular health education materials based on the American Heart Association's Life's Essential 8 framework.
  Interventions: Behavioral: Multidimensional Sleep Health Promotion Intervention
- Standard of care (No Intervention): Participants randomized to the control arm will receive standard American Heart Association Life's Essential 8 cardiovascular health education materials, providing guidance on healthy sleep duration only.

INTERVENTIONS:
Behavioral: Multidimensional Sleep Health Promotion Intervention — Multi-component multidimensional sleep health promotion intervention that includes goal setting, action planning, sleep health coaching and sleep hygiene education, a fixed sleep schedule, self-monitoring, personalized feedback and supportive accountability, and addressing light and noise in the sleep environment.
  Arms: Multidimensional Sleep Health Promotion Intervention

SUMMARY:
The purpose of this randomized clinical trial is to evaluate the impact of a multidimensional sleep health promotion intervention on blood pressure, glycemic control indicators, anthropometric markers of adiposity, and lifestyle factors in adults. Participants will be randomized into an intervention or a control group. The control arm will receive standard Life's Essential 8 cardiovascular health educational materials. The intervention arm will additionally receive a multi-component intervention aimed at improving sleep health based on evidence-based sleep hygiene education and established behavior change techniques that include personalized sleep health feedback, goal setting and establishing a sleep health plan, coaching, self-monitoring, and addressing light and noise in the sleep environment. Mixed methods will be used to understand implementation determinants, processes, and outcomes, ensuring the successful completion and future expansion of this intervention.

DETAILED DESCRIPTION:
Improving multiple domains of cardiometabolic health through contextual behavioral interventions can have far-reaching effects for reducing the burden of multiple cardiometabolic morbidities. Despite a strong evidence base supporting the role of sleep as a major contributor to cardiometabolic health preservation, most lifestyle interventions have targeted diet or physical activity and not sleep. Sleep is amenable to intervention and can improve cardiometabolic health through complementary or synergistic biologic pathways with other lifestyle factors. Therefore, pragmatic multidimensional sleep health interventions may elucidate scalable and sustainable contextual behavioral approaches to improve cardiometabolic health and extend healthspan.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30-65 years
* English or Spanish speaking
* Systolic blood pressure greater than or equal to 120 mmHg
* Sub-optimal sleep health
* No history of overt cardiovascular disease
* No history of cancer

Exclusion Criteria:

* Optimal sleep health
* History of cardiovascular disease or cancer
* Non-English or non-Spanish speaking
* Not cognitively able to complete study requirements
* Severe psychiatric disorders
* Inability to provide informed consent

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in office systolic blood pressure | Baseline, 8 weeks
  The change office systolic blood pressure (mmHg) from baseline to follow-up at 8 weeks will be calculated and compared across randomization arms.

SECONDARY OUTCOMES:
Change in office systolic blood pressure (sustained effect at 24 weeks) | Baseline, 24 weeks
  The change office systolic blood pressure (mmHg) from baseline to follow-up at 24 weeks will be calculated and compared across randomization arms.
Change in office diastolic blood pressure | Baseline, 8 weeks, and 24 weeks
  The change office diastolic blood pressure (mmHg) from baseline to follow-up at 8 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in out-of-office blood pressure | Baseline, 8 weeks, and 24 weeks
  Mean daytime blood pressure (mean of blood pressure readings during the awake period), nighttime blood pressure (mean of blood pressure readings during the asleep period) and mean 24-h blood pressure (mean of the awake and asleep blood pressure values, weighted by the relative amounts of time spent awake and asleep) will be computed using valid readings from ambulatory blood pressure monitoring. Changes in these out-of-office blood pressure metrics from baseline to follow-up at 8 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in fasting glucose | Baseline, 8 weeks, and 24 weeks
  The change in fasting glucose (mg/dl) from baseline to follow-up at 8 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in body weight | Baseline, 8 weeks, and 24 weeks
  The change in body weight (lbs) from baseline to follow-up at 8 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in waist circumference | Baseline, 8 weeks, and 24 weeks
  The change in waist circumference (inches) from baseline to follow-up at 8 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in diet quality | Baseline, 8 weeks, and 24 weeks
  The Mediterranean Eating Pattern for Americans (MEPA) scale, which captures adherence to a heart healthy dietary pattern, will be used to assess diet quality. The MEPA score ranges from 0-16 with higher scores indicating better diet quality. The change in MEPA scores from baseline to 8 weeks and 24 weeks will be calculated and compared across randomization arms.
Change in sleep health | Baseline, 8 weeks, and 24 weeks
  Sleep health will be assessed using sleep duration, regularity, efficiency, and timing from wrist actigraphy and self-reported sleep satisfaction and alertness (measured by daytime sleepiness). Optimal sleep health will be defined as having an average sleep duration (hours/night) ≥7 hours and <9 hours, regular sleep duration and timing (standard deviation of sleep duration and timing variables <90 minutes), sleep efficiency (%) ≥85%, an earlier sleep period (sleep midpoint earlier than 4:00 AM), normal daytime sleepiness (Epworth Sleepiness Scale ≤10), and good self-rated sleep satisfaction and quality. Sleep health will be assessed at baseline, 8 weeks, and 24 weeks. Changes in sleep health from baseline to follow-up at 8 weeks and 24 weeks will be calculated and compared across randomization arms.
Acceptability of Implementation | 8 weeks and 24 weeks
  Acceptability will be measured by questionnaire. Items are adapted from the validated Acceptability of Implementation Measure (AIM) and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better intervention acceptability. The items are analyzed individually and not summed to a total score.
Feasibility of Implementation | 8 weeks and 24 weeks
  Feasibility will be measured by questionnaire using items adapted from the validated Feasibility of Implementation Measure (FIM) and rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better feasibility. The items are analyzed individually and not summed to a total score.
Appropriateness of Implementation | 8 weeks and 24 weeks
  Appropriateness will be measured by questionnaire. Items are adapted from the validated Implementation Appropriateness Measure (IAM) and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better appropriateness. The items are analyzed individually and not summed to a total score.
Satisfaction with intervention | 8 weeks and 24 weeks
  Net promoter score and questions about satisfaction with various intervention components.
Qualitative feedback from interviews on intervention feasibility and implementation | 8 weeks and 24 weeks
  Qualitative feedback on satisfaction, feasibility, acceptability, appropriateness, and scalability will be gathered from participants and staff

CONTACTS AND LOCATIONS:
Overall Officials: Nour Makarem, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, Mailman School of Public Health, New York, New York, United States